CLINICAL TRIAL: NCT01114633
Title: Obesity and Clinical Presentation of Hyperandrogenism
Status: Completed | Type: Observational
Sponsor: Taipei Medical University WanFang Hospital (Other)
Responsible Party: Principal Investigator, Ming-I Hsu, Attending Doctor, Taipei Medical University WanFang Hospital
Other Study IDs: WFH-PCOS-98039
Record Dates: First submitted 2010-04-29; First posted 2010-05-03 (Estimated); Last update posted 2013-11-06 (Estimated); Status verified 2013-11

CONDITIONS: Polycystic Ovary Syndrome
Keywords: PCOS; Acne; Hirsutism
MeSH Terms: conditions — Polycystic Ovary Syndrome; Acne Vulgaris; Hirsutism

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Polycystic Ovarian Syndrome (PCOS) is the most common endocrine disorder in reproductive women. It is estimated that 5 to 10% of women of reproductive age have PCOS. One of the major diagnostic criteria of PCOS was chronic anovulation which lead to irregular menstruation, amenorrhea, and infertility; the other diagnostic criteria was hyperandrogenism which lead to hirsutism, acne and alopecia. Furthermore, PCOS is thought as a metabolic disorder, the long-term consequence of PCOS were diabetes mellitus and cardiovascular disease, which are potentially dangerous in women health. Early diagnosis and prevention is very important to the PCOS patients.

Obesity is the most potential risk of threat to health of populations. There is a major impact of obesity on the PCOS related disorders. Insulin resistance and distribution of adipose tissue were thought to be the important risk factors of cardiovascular and metabolic syndrome. To treat PCOS patients properly,Wan-Fang hospital had established a specific medical team. The investigators recently published in "Fertility and Sterility" about the clinical presentation of androgen excess in Taiwanese women. Hirsutism is much less prevalence (30%) in Taiwanese PCOS women than that previous reported (65-80%) in theWestern women. It is important to know that some clinical presentation of PCOS might have ethic variance. Insulin resistance was reported as another candidate that might have ethic variance. The investigators had reported about 40% women in PCOS women were obese, it is similar with previous literature reported. Obesity is a major factor that could be controlled during the treatment of PCOS.Weight reduction is one of our methods in PCOS treatment. The progressive results for obese PCOS women would be facing the risks of diabetes and metabolic syndrome. The investigators thought like to evaluate the benefit of weight reduction program to the prognosis of obese women with PCOS.

Furthermore, it is known that Endothelial progenitor cells (EPC) be an early marker of cardiovascular disease, the investigators would like to know the role of EPC to predict metabolic syndrome in women with PCOS. Wan-Fang hospital has a professional team in PCOS treatment and research which including gynecological endocrinologist, cardiologist, medical endocrinologist, specialist in weight reduction. This team had been working well for more that 4 years.

The investigators hope that we can make a contribution to the study and treatment of PCOS in Taiwan.

ELIGIBILITY:
Inclusion Criteria:

* Acne and/or hirsutism

Exclusion Criteria:

* Male
* Menopause
* Tumor

Ages: 15 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Polycystic Ovary Syndrome(PCOS)
Sampling Method: Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2009-06; Primary Completion 2010-04 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ming-I Hsu, MD, Principal Investigator — Taipei Medical University WanFang Hospital
Locations (1):
- Taipei Medical University WanFang Hospital, Taipei, Taiwan, Taiwan